CLINICAL TRIAL: NCT02669277
Title: Safety, Tolerability and Efficacy of Single Dose Low Cost Minipool Intravenous Immunoglobulins in Moderately Severe Newly Diagnosed ITP: A Prospective Randomized Study
Brief Title: Safety, Tolerability and Efficacy of Single Dose Low Cost Minipool Intravenous Immunoglobulins in Moderately Severe Newly Diagnosed ITP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohsen Saleh Elalfy, professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU R30/2015
Record Dates: First submitted 2016-01-20; First posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Newly Diagnosed Pediatric ITP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- group A (No Intervention): no platelet enhancing therapy
- group B (Active Comparator): Standard IVIG single dose 1.0 gm /kg/dose
  Interventions: Drug: standard IVIG product
- group C (Experimental): minipool IVIG product single dose 1.0 gm /kg/dose
  Interventions: Drug: IVIG prepared by minipool technology

INTERVENTIONS:
Drug: IVIG prepared by minipool technology — Drug: To demonstrate the efficacy of new product IVIG prepared by minipool technology as assessed by Bleeding Score and platelet count at 3 days, 1 week, 2 weeks and 4 weeks.
  Other Names: IG plasma
  Arms: group C
Drug: standard IVIG product — to compare efficacy and safety with the minipool IVIG
  Arms: group B

SUMMARY:
To demonstrate the efficacy of new product IVIG prepared by minipool technology as assessed by Bleeding Score and platelet count at 3 days, 1 week, 2 weeks and 4 weeks.

The platelet response rate is defined as the percentage of subjects responding to treatment with an increase of platelet count from ≤ 20 x 10^9/L to ≥ 100 x 10^9/L and absence of bleeding (complete response) or platelet count ≥ 50 x 10^9/L and at least 2-fold increase the base line count with absence of bleeding (partial response), within the specified time frame.

DETAILED DESCRIPTION:
To demonstrate the efficacy of new product IVIG prepared by minipool technology as assessed by Bleeding Score and platelet count at 3 days, 1 week, 2 weeks and 4 weeks.

The platelet response rate is defined as the percentage of subjects responding to treatment with an increase of platelet count from ≤ 20 x 10^9/L to ≥ 100 x 10^9/L and absence of bleeding (complete response) or platelet count ≥ 50 x 10^9/L and at least 2-fold increase the base line count with absence of bleeding (partial response), within the specified time frame.

Secondary:

1. To assess safety of mini-pool IVIG in patients with newly diagnosed ITP by assessing frequency of adverse events related to mini-pool IgG administration
2. To compare data on efficacy and safety of mini-pool IVIG with data obtained from literature on standard IVIG.

Study population:

Patients with newly diagnosed ITP attending Hematology clinic Ain Shams Children hospital

Sample size:

Seventy- two patients will be enrolled. They will be divided into 3 groups:

Group A; platelet non enhancing group Group B; group receiving standard IVIG Group C; group receiving IVIG New product 24 patients in each group in a ratio 1:1:1.

ELIGIBILITY:
Inclusion Criteria:

1. All newly diagnosed ITP patients (< 2 weeks from onset of the disease), with no platelet enhancing therapy.
2. Age eligible for study: 1-16 years old
3. Gender eligible for study: both sexes
4. Informed consent signed by patient or his legal guardian.

Exclusion Criteria:

1. Patients started on steroid therapy.
2. Platelet count<10,000/mm3.
3. Having a life threatening bleeding.
4. Patients with known or suspected hypersensitivity to immunoglobulins or previous severe side effects to immunoglobulin therapy.
5. Treatment with immunosuppressive or other immunomodulatory drugs within 3 weeks prior to screening.
6. Treatment with any other investigational drug within 7 days before study entry.

Ages: 12 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
bleeding score(SMOG) | 4 weeks
  change of bleeding score(SMOG) at day 3,week1,week 2 and week 4 after presentation
complete blood count | 4 weeks
  change of complete blood count for number of platelets,absolute neutrophil count,absolute lymphocyte count and hemoglobin at day 3,week 1,week 2 and week 4 after presentation

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 4 weeks
  presence of side effects: anaphylaxis,fever,rash and any others

CONTACTS AND LOCATIONS:
Locations (1):
- hematology clinic ,pediatrics hospital, Ain Shams University hospital Cairo, Egypt, Cairo, Egypt